CLINICAL TRIAL: NCT07348874
Title: Predictive Accuracy of Machine Perfusion Parameters for Kidney Allograft Outcome - A National Analysis Following the Commencement of Hypothermic Machine Preservation of Extended Criteria Donor (ECD) Kidneys in Germany
Brief Title: Predictive Accuracy of Machine Perfusion for Kidney Transplant Outcomes in Germany
Acronym: PRE-MAP-Kidney
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Peri Husen, MD, University Hospital Heidelberg
Record Dates: First submitted 2025-12-30; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant; Renal Transplant; Organ Preservation
Keywords: Machine Perfusion; Hypothermic Machine Perfusion; Upfront Machine Perfusion; Continuous Machine Perfusion; Organ Preservation; Marginal Allograft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Continuous HMP: Patients receiving ECD-DBD kidney allograft after continuous HMP at German Transplant centres

SUMMARY:
Kidney transplantation remains the only definitive treatment for end-stage renal disease, yet the increasing use of extended criteria donor (ECD) kidneys heightens the risk of ischemia-reperfusion injury, particularly under static cold storage (SCS). Continuous hypothermic machine perfusion (HMP) has been introduced to improve preservation quality, but robust clinical evidence regarding its predictive value for post-transplant outcomes in ECD kidneys after donation after brain death (DBD) is limited.

The PRE-MAP Kidney Study is a prospective, non-interventional, multicenter observational study conducted across all German transplant centers. The study systematically collects technical machine perfusion parameters (flow, resistance, perfusion duration) and correlates these with clinical outcomes following kidney transplantation.

The primary endpoint is 12-month kidney function (eGFR). Secondary endpoints include surgical complications, length of stay, and transplant-specific events (acute rejection, primary non-function, delayed graft function).

This national cohort aims to determine the prognostic significance of HMP parameters in marginal donor kidneys and to generate evidence supporting future recommendations for organ preservation and allocation practices.

DETAILED DESCRIPTION:
The PRE-MAP Kidney Study is a prospective, multicenter, observational clinical trial conducted across all German kidney transplant centers following the nationwide introduction of continuous hypothermic machine perfusion (HMP) for extended criteria donor (ECD) kidneys. The primary objective is to evaluate the association between machine perfusion parameters obtained during continuous HMP and post-transplant allograft function, with a specific focus on 12-month kidney function assessed by estimated glomerular filtration rate (eGFR). Secondary objectives include evaluating short- and mid-term transplant outcomes such as delayed graft function (DGF), primary non-function (PNF), biopsy-proven acute rejection, recipient and graft survival, and postoperative clinical course.

Rationale and Background Kidney transplantation is the standard therapy for end-stage renal disease. Due to donor organ scarcity, an increasing proportion of transplanted kidneys meet extended criteria (ECD), making them more susceptible to ischemia-reperfusion injury. Static cold storage (SCS), the conventional preservation method, has been shown to be associated with higher risks of impaired graft function in marginal organs. Continuous HMP has been introduced nationwide in Germany following the 2024 recommendations of the German Medical Association for ECD kidneys, allowing ex-vivo hypothermic perfusion during graft transport and offering the potential to improve organ viability. However, robust clinical data linking perfusion parameters-such as flow, pressure, resistance, temperature, and perfusion duration-to transplant outcomes in real-world practice remain limited. The PRE-MAP Kidney Study addresses this gap by prospectively collecting perfusion and clinical data under routine care conditions without altering allocation or clinical management.

Study Design The study is designed as a prospective, multicenter, non-interventional observational cohort trial. All participating German transplant centers will consecutively enroll eligible recipients of ECD kidneys preserved via continuous HMP. The study does not modify surgical retrieval techniques, organ allocation procedures, or clinical management protocols. Machine perfusion is performed exclusively within the national organ procurement framework of the Deutsche Stiftung Organtransplantation (DSO) using the CE-certified ORS LifePort Kidney Transporter.

Continuous HMP is initiated immediately after organ retrieval in donor hospitals per manufacturer guidelines. Perfusion-specific parameters-including flow, pressure, temperature, and perfusion duration-are automatically recorded throughout transport. Upon arrival at the recipient center, the graft is disconnected from the device and transplanted according to local standards. Postoperative and outpatient follow-up follow standard institutional routines without additional study-specific interventions. All patients are followed for 12 months post-transplantation.

Endpoints Primary Endpoint Kidney function at 12 months post-transplantation assessed by eGFR.

Secondary Endpoints Recipient and graft survival at 12 months Kidney function at 3 and 6 months (eGFR) Incidence of delayed graft function (DGF), defined as dialysis within the first post-transplant week Incidence of functional DGF (<10% serum creatinine decrease over 3 consecutive days in the first week) Primary non-function (dialysis requirement at 3 months) Total organ preservation time Incidence of biopsy-proven acute rejection

Patient Population Eligible participants are adult kidney transplant candidates listed at Eurotransplant who receive an ECD kidney donor allograft from donation after brain death (DBD). ECD criteria follow international definitions: donor age ≥60 years, or donor age 50-59 years with two of the following-cerebrovascular cause of death, history of hypertension, or terminal serum creatinine >1.5 mg/dL. Recipients must provide written informed consent upon admission to the transplant center. Exclusion criteria include living donor transplantation, combined organ transplantation, participation in interventional trials affecting outcomes, inability to comply with study requirements, or language barriers.

Study Procedures The study does not alter organ allocation, retrieval, transplantation, or postoperative care. Organ retrieval is performed by trained DSO surgical teams. Device connection and perfusion setup are carried out by certified procurement surgeons and perfusionists. Continuous HMP is applied exclusively during ex-vivo transport. Upon arrival, transplantation proceeds according to local practice. Follow-up examinations occur within routine outpatient visits. Clinical and perfusion data are documented pseudonymously in standardized case report forms (CRFs).

Statistical Analysis The primary endpoint (12-month eGFR) will be analyzed using multivariable linear regression to evaluate associations with HMP perfusion parameters, adjusted for relevant donor, recipient, and procedural factors. Secondary endpoints will be assessed using appropriate statistical methods, including non-parametric tests, ANCOVA models, logistic regression, Cox proportional hazards models, and descriptive analyses. Continuous variables will be summarized by mean, median, and distribution; categorical variables by frequency and percentage. All tests will be two-sided with a significance threshold of 0.05.

Ethical Conduct and Data Protection The study is conducted in accordance with the Declaration of Helsinki, ICH-GCP principles, and German regulatory requirements. Institutional Review Board (IRB) approval will be obtained prior to initiation. All participants provide informed consent. Data are pseudonymized and shared only with authorized parties in compliance with data protection regulations. The device used in the study is CE-certified and applied strictly within its intended use without adding risks or burdens for recipients.

Study Duration and Timeline The recruitment phase is planned to begin in January 2026 following the first implementation of continuous HMP within the DSO network, and will continue for approximately 12 months. Each participant is followed for 12 months post-transplantation. Including data evaluation and final reporting, total study duration is approximately 26 months.

Safety Considerations Because this is a non-interventional observational study involving a CE-certified medical device used according to standard practice, no study-specific safety risks are anticipated. No additional diagnostic or therapeutic procedures are required. Study termination would occur only for administrative or organizational reasons.

Post-Study Care After study completion, participants return fully to routine clinical care. No additional treatment is required as a consequence of study participation, and withdrawal does not affect access to standard medical care.

Infrastructure The study is conducted at all German kidney transplant centers in collaboration with the DSO network. ORS LifePort Kidney Transporter devices are available for continuous use throughout the study period. Principal investigators and participating teams have extensive clinical and research experience in organ transplantation and machine perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patients 18 years or older
3. Listed for kidney transplantation (KT)
4. Receiving ECD* donation after brain death kidney allografts following national organ procurement
5. Kidney allograft being transported at continuous HMP
6. Transplantation of recipient at a national transplant center

   * Extended Criteria Donation:

1. Donor age ≥ 60 years 2. Donor age 50 - 59 plus 2 additional attributes: I. Arterial hypertension in medical history II. Last serum creatinine >1.5mg/dL (133mmol/L) III. Cerebrovascular cause of death

Exclusion Criteria:

1. Recipients of living donor KT
2. Combined transplantations (liver-kidney, kidney-pancreas, etc.)
3. Participation in another intervention-trial with interference of intervention and/or outcome of this study
4. Unwilling or unable to follow the procedures outlined in the protocol
5. Mentally or legally incapacitated
6. Inability to understand the procedures due to language barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients waitlisted at a German transplant center for kidney transplantation receiving an ECD donor allograft from donation after brain death after continuous hypothermic oxygenated machine perfusion
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2028-01-19 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Kidney Function | 1 year after kidney transplantation
  Kidney function assessed by the estimated glomerular filtration rate

SECONDARY OUTCOMES:
Recipient and graft survival | 1 year after kidney transplantation
  Recipient graft survival
Kidney function | 1, 3 and 6 months after kidney transplantation
  Kidney function assessed by estimated glomerular filtration rate (eGFR)
Delayed Graft Function (DGF) | 7 days after kidney transplantation
  Incidence of delayed graft function (requirement of dialysis during the first week following kidney transplantation with return of kidney function)
Primary Non-Function | 3 months after kidney transplantation
  Primary non-function (PNF): patient requires dialysis at 3 months after kidney transplantation
Total organ preservation of the donor kidney | From placement of the donor kidney to the machine perfusion device until removal of the donor kidney from the machine perfusion device (measured in minutes)
  Total organ preservation time of the donor kidney
Acute rejection episodes | From enrollment until the end of follow up at 1 year post kidney transplantation
  Incidence of biopsy proven acute rejection episodes

IPD SHARING:
Plan to Share IPD: Undecided